CLINICAL TRIAL: NCT04731480
Title: Evaluation of Propofol Total Intravenous Anaesthesia Administered by Closed Loop Anaesthesia Delivery System Versus Target Controlled Infusion Device in Adults Undergoing Non-Cardiac Surgery: A Randomised Controlled Study
Brief Title: Comparison of TIVA by Closed Loop Anaesthesia Delivery System Versus Target Controlled Infusion Device
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sir Ganga Ram Hospital (Other)
Responsible Party: Principal Investigator, Nitin Sethi, DNB, Senior Consultant, Sir Ganga Ram Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: EC/12/20/1787
Record Dates: First submitted 2021-01-25; First posted 2021-02-01 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Anesthesia
MeSH Terms: interventions — Propofol

STUDY DESIGN:
Intervention Model Description: One hundred sixty-participants (40/group) aged 18-65 years, ASA physical status I-II, of either sex, and undergoing elective non-cardiac surgery of minimum 60-minutes duration recruitment will be randomly divided into one of the four groups:
  Group-1 [CLADS group, n= 40, study group], Group-2 [Marsh model (MM) group, n= 40, study group], Group-3 [Schneider Model (SM) Group, n= 40, study group], and Group-4 [Manual (M) Group, n= 40, Control group].
Who Masked: Participant, Outcomes Assessor
Masking Description: Inside the operating, the attending anaesthesiologist will not be blinded to the technique utilized to administer general anaesthesia (GA) and the recovery parameters immediately after extubation. However, the postoperative patient recovery profile will be evaluated by an independent assessor blinded to the GA technique and peri-extubation profile.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- CLADS group (Active Comparator): Propofol administration rate will be controlled by a feedback loop facilitated by BIS monitoring using the closed-loop anaesthesia delivery system (CLADS). A BIS value of 50 will be used as the target point for induction and maintenance of anesthesia.
  Interventions: Drug: Propofol
- Marsh model group (Active Comparator): The target-controlled infusion (TCI) pump will be programmed to marsh model with the target plasma site concentration of 3-µg/ml. The plasma concentration will be altered to maintain a target BIS of 50 during induction and maintenance of anesthesia
  Interventions: Drug: Propofol
- Schnider model group (Active Comparator): The TCI-pump will be programmed to will be programmed to Schnider model with the target effect site concentration of 3-µg/ml. The effect-site concentration will be altered to maintain a target BIS of 50 during induction and maintenance of anesthesia.
  Interventions: Drug: Propofol
- Manual group (Active Comparator): Propofol administration will be controlled manually using an intravenous infusion pump to maintain a target BIS of 50 during induction and maintenance of anesthesia.
  Interventions: Drug: Propofol

INTERVENTIONS:
Drug: Propofol — Propofol administration rate will be controlled by a feedback loop facilitated by BIS monitoring using the closed loop anaesthesia delivery system (CLADS). A BIS value of 50 will be used as the target point for induction and maintenance of anaesthesia.
  Arms: CLADS group
Drug: Propofol — The target controlled infusion (TCI) pump will be programmed to marsh model with the target plasma site concentration of 3-µg/ml. The plasma concentration will be altered to maintain a target BIS of 50 during induction and maintenance of anesthesia
  Arms: Marsh model group
Drug: Propofol — The target controlled infusion (TCI) pump will be programmed to Schneider model with the target effect site concentration of 3-µg/ml. The effect-site concentration will be altered to maintain a target BIS of 50 during induction and maintenance of anesthesia
  Arms: Schnider model group
Drug: Propofol — Manual propofol administration will be done using an intravenous infusion pump to maintain a target BIS of 50 during induction and maintenance of anesthesia.
  Arms: Manual group

SUMMARY:
Total intravenous anaesthesia (TIVA) is now being adopted as a preferred technique for providing GA because of its various inherent advantages like reduced PONV incidence, improved quality of recovery post GA, anti-inflammatory and anti-oxidant action, anti-neoplastic activity, analgesic action, and absence of greenhouse effect. Over the years propofol-TIVA delivery has become more methodical due to the use of target-controlled infusion (TCI) systems. The current TCI technology has evolved with the introduction of the 'open' TCI concept wherein syringes of any configuration can be attached to the TCI-pumps having pre-programmed propofol PK-PD models. The two most commonly use propofol PK-PD models are the Marsh and Schneider models targeting the propofol blood plasma concentration and effect site concentration in the brain respectively. Automated delivery of propofol using computer-controlled closed loop anaesthesia device delivers propofol based on patient's frontal cortex electrical activity as determined by bispectral index (BIS). Evaluation of anaesthesia delivery by these systems has shown that they deliver propofol and maintain depth of anaesthesia with far more precision as compared to manual administration. A recent advance in propofol delivery has been the development of automated closed loop anaesthesia delivery system. These devices deliver propofol based on patient's frontal cortex electrical activity as determined by bispectral index (BIS).Closed loop anaesthesia delivery system (CLADS) is an indigenously developed continuous automated intravenous infusion system which delivers propofol based on patients' EEG profile (BIS) feedback. Currently there is no data available comparing the efficacy of TCI delivered propofol versus automated propofol delivery systems. The investigators hypothesize that automated propofol delivery by CLADS will provide more consistent anaesthesia depth maintenance as compared to TCI delivered propofol. This randomized controlled study aims to compare the efficiency of CLADS-driven propofol TIVA versus TCI administered in patients undergoing non-cardiac surgery with respect to adequacy of anaesthesia depth maintenance, performance characteristic of propofol delivery system hemodynamic stability, recovery from anaesthesia and postoperative sedation.

DETAILED DESCRIPTION:
Inhalation anaesthetic were backbone of general anaesthesia (GA) practice till the time an intravenous anaesthetic, propofol was introduced in early 1970's and its commercial availability in 1980's, which led to the resurgence in the practice of total intravenous anaesthesia (TIVA). TIVA is now being adopted as a preferred technique for providing GA because of scores of inherent advantages, like, reduced PONV incidence, improved quality of post-anaesthesia recovery, anti-inflammatory and anti-oxidant action, anti-neoplastic activity, analgesic action, and absence of greenhouse effect among many others.Over the years propofol-TIVA delivery has become more methodical and precise owing to the use of target controlled infusion (TCI) systems. TCI systems use propofol pharmacokinetic (PK) or pharmacodynamics (PD) models which predict either the plasma or the effect-site propofol concentration required for maintenance of GA steady-state during surgery. The 'Diprifusor' TCI-system was the first commercially available propofol TCI-system. The 'Diprifusor' TCI-system was a 'closed' TCI-system which required a special electronically tagged pre-filled propofol syringe to be attached to the TCI-pump. The current TCI technology has evolved with the introduction of the 'open' TCI concept wherein syringes of any configuration can be attached to the TCI-pumps having pre-programmed propofol PK-PD models. Currently, the two most commonly used PK-PD models that drive TCI systems to deliver TIVA are the 'Marsh' and 'Schneider' models. Whereas Marsh model targets blood plasma concentration of propofol for anaesthesia maintenance, the Schneider model targets effect-site concentration in the brain. A recent advance in propofol TIVA delivery has been the development of automated closed loop anaesthesia delivery system. These devices deliver propofol based ascertaining patient's frontal cortex electrical activity as determined by bispectral index (BIS) score and then keeping the values within a pre-assigned range consistent with robust GA depth. Closed loop anaesthesia delivery system (CLADS) is an indigenously developed patented (502/DEL/2003) computer-controlled anaesthesia delivery system. CLADS typically works with feedback loop information elicited by BIS monitoring and delivers propofol TIVA to the patient via a non-TCI automated infusion pump. This basis of CLADS is the control algorithm based on the relationship between diverse rates of propofol infusion and the processed EEG variable. Although propofol delivery by CLADS is based on pharmacokinetic model but for greater precision and efficient administration, its delivery trigger is directly linked with feedback mechanism involving patient's EEG profile as monitored by the BIS scores. In a multicentre study on evaluation of anaesthesia delivery by CLADS, it was shown that CLADS maintains depth of anaesthesia with far more precision as compared to manual administration. Queerly while TCI & CLADS technology evolved over a period of time; there is no data available comparing the efficacy of TCI delivered propofol-TIVA versus automated propofol delivery systems. Based on additional feedback loop incorporated to the PK-PD model the investigators contend that automated propofol TIVA as administered by CLADS is likely to be superior to TCI system in achieving and sustaining anaesthesia depth. This randomized controlled study aims to compare the efficacy of CLADS-driven propofol TIVA versus TCI administered propofol TIVA in adult patients undergoing non-cardiac surgery with respect to: adequacy of anaesthesia depth maintenance (primary objective), performance characteristic of propofol delivery system, propofol requirement, hemodynamic stability, recovery from anaesthesia and postoperative sedation (secondary objectives).

ELIGIBILITY:
Inclusion Criteria:

* aged 18-65 years
* ASA physical status I-II
* undergoing elective non-cardiac surgery of minimum 60-minutes duration

Exclusion Criteria:

* Uncompensated cardiovascular disease (e.g. uncontrolled hypertension, atrio-ventricular block, sinus bradycardia, congenital heart disease, reduced LV compliance, diastolic dysfunction)
* Hepato-renal insufficiency
* Uncontrolled endocrinology disease (e.g. diabetes mellitus, hypothyroidism)
* Known allergy/hypersensitivity to the study drug
* Drug dependence/substance abuse
* Requirement of postoperative ventilation
* Refusal to informed consent

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2021-02-02 (Actual); Primary Completion 2025-06-17 (Actual); Study Completion 2025-06-17 (Actual)

PRIMARY OUTCOMES:
Anaesthesia depth consistency | From end of surgery till 8 hours intraoperatively
  It will be determined by the percentage of the anaesthesia time during which the BIS remained +/- 10 of the target BIS of 50

SECONDARY OUTCOMES:
Performance characteristic of propofol delivery system | From end of surgery till 10-hours intraoperatively
  It will be determined using the Varvel criteria parameter :median performance error (MDPE). This parameter is calculated by the computer software which analyses the intraoperative BIS data. This parameter have no unit of measurement. Its just a abstract number.
Performance characteristic of propofol delivery system | From end of surgery till 10-hours intraoperatively
  It will be determined using the Varvel criteria parameter: median absolute performance error (MDAPE).This parameter is calculated by the computer software which analyses the intraoperative BIS data. This parameter have no unit of measurement. Its just a abstract number.
Performance characteristic of propofol delivery system | From end of surgery till 10-hours intraoperatively
  It will be determined using the Varvel criteria parameter: wobble. This parameter is calculated by the computer software which analyses the intraoperative BIS data. This parameter have no unit of measurement. Its just a abstract number..
Performance characteristic of propofol delivery system | From end of surgery till 10-hours intraoperatively
  It will be determined using the Varvel criteria parameter: global score. It is calculated using the formula Median absolute performance error + wobble / percentage of the anesthesia time during which the BIS remained +/- 10 of the target BIS of 50. This parameter have no unit of measurement. Its just a abstract number..
Propofol induction dose (mg/kg) | From start of propofol injection till 2-minutes intraoperatively
  Dose of propofol required for induction of anaesthesia
Propofol maintenance dose (mg/kg/hr) | From 2-minutes intraoperatively till 10-hours intraoperatively
  Dose of propofol required for maintenance of anaesthesia
Intra-operative heart Rate (beats per minute) | From beginning of anaesthesia till 10 hours intraoperatively
  Comparison of intra-operative heart rate between the study arms will be done
Intra-operative systolic , diastolic, and mean blood pressure (mmHg) | From beginning of anaesthesia till 10 hours intraoperatively
  Comparison of intra-operative blood pressure- systolic, diastolic, and mean blood pressure between the study arms will be done
Early recovery from anaesthesia | From end of anaesthesia till 20-minutes postoperatively
  Time taken by the patient to open his/her eyes after discontinuation of anaesthesia will be noted
Early recovery from anaesthesia | From end of anaesthesia till 20-minutes postoperatively
  Time taken for tracheal extubation after discontinuation of anaesthesia will be noted
Postoperative sedation | From end of anaesthesia till 24-hours postoperatively
  Will be assessed using Modified Observer's assessment of alertness/sedation scale. The scale has a maximum value of '5', which refers to a fully awake patient and a minimum value of '0' which refers to a deeply sedated patient.
Induction Time | From beginning of anesthesia till 5-minutes intraoperatively
  Time taken for for induction of anesthesia i.e. time taken from starting propofol infusion till a target BIS value of 50 is achieved

CONTACTS AND LOCATIONS:
Overall Officials: Jayashree Sood, MBBS, MD, FFRCA, PGDHHM, FICA, Study Chair — Sir Ganga Ram Hospital, New Delhi, INDIA; Goverdhan D Puri, MBBS, MD, PhD, Study Director — Postgraduate Institute for Medical Education & Research, Chandigarh, India; Nitin Sethi, MBBS, DNB, Principal Investigator — Sir Ganga Ram Hospital, New Delhi, INDIA; Amitabh Dutta, MBBS, MD, PGDHR, Principal Investigator — Sir Ganga Ram Hospital, New Delhi, INDIA
Locations (2):
- India (2):
  - Nitin Sethi, New Delhi, National Capital Territory of Delhi
  - Sir Ganga Ram Hospital, New Delhi, National Capital Territory of Delhi

IPD SHARING:
Plan to Share IPD: No